CLINICAL TRIAL: NCT00926276
Title: The Role of Anti-Reflux Surgery for Gastroesophageal Reflux Disease in Premature Infants With Bronchopulmonary Dysplasia (BPD).
Brief Title: The Role of Anti-Reflux Surgery for Gastroesophageal Reflux Disease in Premature Infants With Bronchopulmonary Dysplasia
Acronym: GERD-BPD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, KuoJen Tsao, Assistant Professor - Pediatric Surgery, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GERD-BPD
Record Dates: First submitted 2009-06-19; First posted 2009-06-23 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Gastroesophageal Reflux Disease; Bronchopulmonary Dysplasia
Keywords: Gastroesophageal Reflux Disease (GERD); Bronchopulmonary Dysplasia (BPD); Fundoplication
MeSH Terms: conditions — Gastroesophageal Reflux; Bronchopulmonary Dysplasia | interventions — Fundoplication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Surgical Treatment Group-Fundoplication (Active Comparator): Re-evaluated 1 month post-op Re-evaluated 2 months post-op
  Interventions: Procedure: Fundoplication
- Medical Therapy (Active Comparator): Treated by primary clinician for GERD Re-evaluated 1 month Proceed to Fundoplication if GERD persist by pH-MII Re-evaluated at 2 months (1 month post-op) Worsening BPD will be given option of immediate surgery
  Interventions: Procedure: Fundoplication

INTERVENTIONS:
Procedure: Fundoplication — Fundoplication

SUMMARY:
The purpose of this study is to evaluate the efficacy of fundoplication in premature infants with GERD and BPD.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) has been postulated to result in chronic aspiration contributing to the development of chronic lung disease, otherwise known as bronchopulmonary dysplasia (BPD) in premature infants. This association has been indirectly based on anecdotal improvement in the respiratory status of infants with BPD after anti-reflux therapy, but the direct causal relationship has been difficult to prove. In addition, the historical evidence for infants with GERD has been based on acid reflux only which is diagnosed by 24 hour intra-esophageal pH monitoring, the gold standard. However, with the introduction of multi-channel intraluminal impedance (MII), GERD can now include non-acid reflux. The contribution of non-acid reflux to the development of BPD in premature infants is unknown. As our understanding of GERD has improved, previous assumptions regarding the efficacy of therapy may no longer be valid. The utilization of anti-reflux surgery (fundoplication) for the treatment of BPD in premature infants with GERD has not been rigorously studied. The efficacy of fundoplication in this patient population has yet to be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Must meet all inclusion criteria for Initial Evaluation of GERD
2. Positive pH-MII test for GERD
3. Upper GI contrast radiograph to evaluate for associated congenital gastrointestinal anomalies
4. > or = 2 kg (due to technical limitations of fundoplication)

Exclusion Criteria:

1. Previous intra-abdominal surgery except for gastrostomy
2. Those deemed not surgical candidates
3. Infants with associated congenital gastrointestinal anomalies
4. > or = 1 year of age at time of Initial Evaluation of GERD

Ages: 24 Weeks to 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 2 (Actual)
Dates: Start 2009-06; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of fundoplication in premature infants with GERD and BPD. | Three months

SECONDARY OUTCOMES:
Establish preliminary data regarding the correlation between acid and non-acid GERD and pepsin from tracheal aspirates as a marker of chronic aspiration in premature infants with BPD. | Six months

CONTACTS AND LOCATIONS:
Overall Officials: KuoJen Tsao, M.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- UT-Houston Pediatric Surgery & Memorial Hermann Children's Hospital, Houston, Texas, United States